CLINICAL TRIAL: NCT03100864
Title: Exploratory Trial to Assess Mechanism of Action, Clinical Effect, Safety and Tolerability of 12 Weeks of Treatment With BI 655130 in Patients With Active Ulcerative Colitis (UC)
Brief Title: This Study Tests How BI 655130 Works in Patients With Active Ulcerative Colitis. The Study Also Tests How Well BI 655130 is Tolerated and Whether it Helps the Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1368-0004; 2017-000100-20 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-04 (Actual); Results first posted 2020-11-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — spesolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spesolimab (Experimental)
  Interventions: Drug: Spesolimab

INTERVENTIONS:
Drug: Spesolimab — 12 weeks treatment

SUMMARY:
The primary objective of this trial is to understand the mechanism of action of BI655130 in patients with UC

Secondary objectives are to explore clinical effect, safety and tolerability (including immunogenicity) of BI 655130 treatment

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years at screening
* Diagnosis of UC >= 3 months prior to screening.
* Moderately to severely active UC as confirmed by Mayo Score ≥6
* Receiving conventional, non-biologic therapy for UC.
* Negative colon cancer screening
* Further inclusion criteria apply

Exclusion Criteria:

* Prior use of any biological treatment in the past (e.g.integrin inhibitors, IL12/23 or IL23 inhibitors, any investigational biological drugs)
* Extensive colonic resection
* Evidence of infection with C. difficile or other intestinal pathogen < 30 days prior to screening
* Active or latent tuberculosis
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- UZ Leuven, Leuven, Belgium
- Germany (2):
  - Asklepios Kliniken Westklinikum Hamburg, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
- Addenbrooke's Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an Phase IIa multi-centre, non-randomised, uncontrolled single arm), open-label, exploratory trial to assess biomarker changes in response to Interleukin-36 signalling blockade induced by treatment with spesolimab in patients with moderate to severe active Ulcerative colitis.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Spesolimab 1200 mg Intravenous (i.v.): 1200 milligram Spesolimab (infusion solution, BI 655130) was given for 12 weeks intravenously with a concentration of 20 milligram/milliliter every four weeks (on Day 1, Week 4, and Week 8).
Period: Overall Study
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): patients who received at least 1 dose of study drug, who had a baseline and at least 1 post baseline measurement for any clinical efficacy or biomarker endpoint without any Important protocol deviation flagged for exclusion or rescue use on or after Visit 1b but prior to administration of the first dose of spesolimab.
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (19.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Total Number of Deregulated Genes Comparing Baseline to Post Treatment, Analysed by Gene Expression of Mucosal Biopsies Via RNA Sequencing, Per Time Point up to Week 12
Description: The total number of deregulated genes comparing baseline to post treatment, analysed by gene expression of mucosal biopsies via RNA sequencing, per time point up to Week 12. A total of 60,675 genes were evaluated, 40,586 genes were included in the differential expression analyses. Based on the raw read count values the DESeq2 method, one of the standard methods to analyse RNAseq data, was used for the gene expression analysis and to identify deregulated genes. A gene was considered deregulated with a FDR (false discovery rate) adjusted p-value < 0.01 and a fold change ≤ -1.3 or ≥ 1.3.
Time Frame: Measurements done at baseline (day -8 to -6), day 1, day 4, day 15, day 57 and day 85 (week 12).
Population: Completers analysis set: completed the trial medication through to end of trial visit, had a baseline and at least 1 post baseline measurement for any clinical efficacy or biomarker endpoint without any Important protocol deviation flagged for exclusion or rescue use on or after Visit 1b but prior to administration of the first dose of spesolimab.
Measure: Number; unit: deregulated genes
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
Number analyzed (Participants) | 5
deregulated genes
  Change from baseline to Day 1 | 3
  Change from baseline to Day 4 | 5
  Change from baseline to Day 15 (week 2) | 2
  Change from baseline to Day 57 (week 8) | 7
  Change from baseline to Day 85 (week 12) | 9

2. Secondary Outcome: Percent Change in C-reactive Protein (CRP) From Baseline to Week 12
Description: Percent change in C-reactive protein (CRP) from baseline to Week 12 (day 85).
Time Frame: Measurements done at baseline (day -8 to -6) and week 12 (day 85).
Population: Safety analysis set (SAF): This patient set included all entered patients who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: percentage change (%)
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
Number analyzed (Participants) | 5
percentage change (%) | -79.6 [-97.9 to 936.7]

3. Secondary Outcome: Percent Change in Faecal Calprotectin From Baseline to Week 12
Description: Percent change in faecal calprotectin from baseline to week 12 (day 85).
Time Frame: Measurements done at baseline (day -8 to -6) and week 12 (day 85).
Population: Safety analysis set (SAF): This patient set included all entered patients who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: percentage change (%)
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
Number analyzed (Participants) | 5
percentage change (%) | 13.0 [-98.7 to 219.3]

4. Secondary Outcome: Percent Change in Faecal Lactoferrin From Baseline to Week 12
Description: Percent change in faecal lactoferrin from baseline to week 12 (day 85).
Time Frame: Measurements done at baseline (day -8 to -6) and week 12 (day 85).
Population: Safety analysis set (SAF): This patient set included all entered patients who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: percentage change (%)
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
Number analyzed (Participants) | 5
percentage change (%) | 0.4 [-99.7 to 388.7]

5. Secondary Outcome: Number of Participants With Clinical Remission (Defined as Mayo Score ≤2 Points, and All Subscores ≤1 Point) at Week 12
Description: Number of participants with clinical remission (defined as Mayo score ≤2 points, and all subscores ≤1 point) at Week 12. The Mayo score is a composite disease activity score consisting of 4 items or subscores: stool frequency (relative to normal), rectal bleeding, physician's global assessment (PGA), and endoscopic appearance. The overall range of the Mayo score was 0 to 12 (higher scores being worse) and each subscore had a range of 0 to 3.
Time Frame: Week 12 (day 85) following start of treatment.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
Number analyzed (Participants) | 5
Participants | 0 [0.000 to 0.434]

6. Secondary Outcome: Number of Patients With Drug Related Adverse Events (AEs)
Description: Number of patients with drug related adverse events (AEs) during the on-treatment period.
Time Frame: Date of start of infusion of first study drug (Day 1) till the date of end of infusion of last study drug (day 57) + 140 days at 11:59 p.m., up to 197 days.
Population: Safety analysis set (SAF): This patient set included all entered patients who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
Number analyzed (Participants) | 8
Participants | 6

ADVERSE EVENTS:
Time Frame: Date of start of infusion of first study drug (Day 1) till the date of end of infusion of last study drug (day 57) + 140 days at 11:59 p.m., up to 197 days.
Description: Safety analysis set (SAF): This patient set included all entered patients who received at least 1 dose of study drug.
Arm/Group | Spesolimab 1200 mg Intravenous (i.v.)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab 1200 mg Intravenous (i.v.) (N=8)
Colitis (Gastrointestinal disorders) | 1
Diverticulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab 1200 mg Intravenous (i.v.) (N=8)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Eye inflammation (Eye disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Gastrointestinal infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 1
Amylase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT03100864/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03100864/SAP_001.pdf